CLINICAL TRIAL: NCT04301362
Title: FIIT Project - Biomarkers of Thrombosis as Predictors of Venous Thromboembolism Risk in Cancer Patients
Brief Title: Biomarkers of Thrombosis as Predictors of Venous Thromboembolism Risk in Cancer Patients
Acronym: FIIT_Score
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centro Hospitalar de Vila Nova de Gaia/Espinho, E.P.E. (Other Government)
Collaborators: LEO Pharma (Industry); Diagnostica Stago (Industry)
Responsible Party: Principal Investigator, Dr. David Ferreira, MD Immunohemotherapy Department, Centro Hospitalar de Vila Nova de Gaia/Espinho, E.P.E.
Other Study IDs: FIIT_Project
Record Dates: First submitted 2020-03-06; First posted 2020-03-10 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Cancer; Thromboembolism; Thrombosis; Biomarkers
Keywords: Khorana; Thrombin generation; Venous thromboembolism
MeSH Terms: conditions — Neoplasms; Thromboembolism; Thrombosis; Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Thrombosis biomarkers — Blood samples shall be prepared according to the manufacturer's instructions and stored at -80°C until analysis. Thrombin generation will be measured using the commercial kit STG®-Tromboscreen kit (Stago). The D-dimers will be quantified using STA LIATEST® D-DI PLUS (Stago).

SUMMARY:
The main venous thromboembolism (VTE) risk prediction model for ambulatory cancer patients is Khorana. Cancer thrombosis is associated with elevated thrombin generation. Its quantification is a promising method for evaluating patient's thrombotic profile.

This study aims to develop a predictive model of VTE risk in ambulatory cancer patients, combining thrombosis biomarkers (D-dimers and thrombin generation potential) with the Khorana score.

This is a prospective observational study that includes newly diagnosed cancer patients proposed for anti-tumor treatment (chemotherapy, immunotherapy or targeted therapies). Patients with disease progression are allowed if chemotherapy-free for 3 months. A 6-month mean incidence of VTE 6-10% is expected, requiring a sample size of 600 patients. Blood sample is collected at inclusion to analyze thrombosis biomarkers and blood count. The primary endpoint is the occurrence of symptomatic or incidental VTE within 6 months of inclusion. Models will follow a logistic approach with K-fold cross-validation (k=10). Model quality will be assessed with Akaike Information Criterion (AIC) and Bayesian Information Criterion (BIC). Decision for entering predictors in multivariate models will be based on p <.10 in the univariate analysis.

DETAILED DESCRIPTION:
The main aims will be the following:

* Evaluate the utility of the combination of thrombosis biomarkers (D-dimers and thrombin generation potential) with the Khorana score in order to stratify VTE risk in ambulatory cancer patients;
* Determine the potential of this new score in the stratification of cancer patients into high- and low-risk VTE groups, in order to identify patients who would benefit from primary thromboprophylaxis;
* Determine the applicability of the thrombin generation test as an independent factor in the stratification of VTE risk in the cancer population under study;
* Determine the predictive value of D-dimers in the cancer population under study (high versus low risk discrimination).

ELIGIBILITY:
Inclusion Criteria:

* Patients older than 18 years.
* Newly diagnosed cancer patients, proposed for anti-tumor medical treatment (chemotherapy, immunotherapy and targeted therapies).
* Patients with a cancer diagnosis, previously under medical anti-tumor treatments, with disease progression proposed for a new line of anti-tumor treatment, who have not recently received chemotherapy (within the last three months).
* Follow-up in Medical Oncology, Clinical Hematology, and Pulmonology consultations at Centro Hospitalar Vila Nova de Gaia/Espinho.

Exclusion Criteria:

* Major bleeding in the last 3 months.
* Major surgery in the last 28 days.
* Patients on anticoagulation/antithrombotic therapy
* Pregnant or breastfeeding women.
* Patients previously submitted to bone marrow transplantation.
* Inaccessibility to the results of the biomarkers or other elements provided for in the Khorana score.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Cancer patients admitted to Medical Oncology, Clinical Hematology, and Pulmonology consultations at Centro Hospitalar Vila Nova de Gaia/Espinho, Portugal.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2019-07-19 (Actual); Primary Completion 2021-07-19 (Estimated); Study Completion 2021-12-19 (Estimated)

PRIMARY OUTCOMES:
Occurrence of symptomatic or incidental VTE | 6 months
  Confirmed by vascular ultrasound, thoracic angiography, and/or ventilation/perfusion scintigraphy. There will be no routine screening for VTE diagnosis. The symptomatic and incidental episodes documented in the clinical process and complementary diagnostic tests will be considered.

SECONDARY OUTCOMES:
Mortality | 6 months
  deaths per 100 persons
Risk factors for the development of VTE | 6 months
  Identify risk factors for the development of VTE in ambulatory cancer patients
Major Bleeding | 6 months
  major bleeding event

CONTACTS AND LOCATIONS:
Overall Officials: David Ferreira, MD, Principal Investigator — Centro Hospitalar Vila Nova de Gaia/Espinho
Locations (1):
- Centro Hospitalar Vila Nova de Gaia/Espinho, Vila Nova de Gaia, Portugal

IPD SHARING:
Plan to Share IPD: No
No applicable